CLINICAL TRIAL: NCT03730324
Title: Developing a Multivariable Diagnostic Prediction Model for Prostate Biopsy Outcome Using Biomarkers and mpMRI as Prediction Variables in Biopsy naïve Men.
Brief Title: Predicting Prostate Biopsy Results With Biomarkers and mpMRI.
Acronym: ProBioM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torben Brøchner Pedersen (Other)
Responsible Party: Sponsor-Investigator, Torben Brøchner Pedersen, PhD-Student, MD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20170043
Record Dates: First submitted 2018-08-21; First posted 2018-11-05 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: Biomarkers; Magnetic Resonance Imaging; Diagnostic
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Multiparametric Magnetic Resonance Imaging; Urination

STUDY DESIGN:
Intervention Model Description: Study subjects will be randomized in a 1:7 fashion between
  1. Standard biopsies + biomarkers and
  2. Biomarkers + mpMRI and Standard / mpMRI targeted biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Study subject will undergo sampling of plasma and urine biomarkers.
  Interventions: Diagnostic Test: Urine and plasma biomarkes.
- Magnetic Resonance Imaging. (Experimental): Prior to biopsies a magnetic resonance imaging scan will be performed.
  Interventions: Diagnostic Test: mpMRI; Diagnostic Test: Urine and plasma biomarkes.

INTERVENTIONS:
Diagnostic Test: mpMRI — Study subjects will undergo urine and plasma biomarker testing and mpMRI prior to biopsy
  Arms: Magnetic Resonance Imaging.
Diagnostic Test: Urine and plasma biomarkes. — Study subjects will undergo urine and plasma biomarker testing prior to standard biopsy

SUMMARY:
Current standard prostate biopsy techniques, used to definitively diagnose prostate cancer (PC), utilises an ultrasound guided biopsy approach, that offers unsatisfactory specificity and sensitivity for clinical significant PC. This often leads to harmful unnecessary biopsies. To improve the overall detection of clinical significant PC, multiparametric magnetic resonance imaging (mpMRI) has emerged as a new technique that might be useful in selecting the appropriate patient for biopsy. Nevertheless, mpMRI fail to detect cancer in some circumstances and the exact role of mpMRI is undetermined. Currently, the majority of PC is diagnosed either incidentally or by unsystematic screening with prostate specific antigen (PSA). PSA suffers from being an organ specific, but cancer unspecific serum biomarker. PSA testing may neither rule out or confirm the presence of prostate cancer. Newer biomarkers have shown promise in curbing some of this sensitivity and specificity gap, but still needs refinement.

In the present study, the investigators will use mpMRI and a new set of urine and plasma biomarkers in combination, prior to performing standard biopsies in order to develop a prediction model for the biopsy outcome. If proven successful the model would offer excellent risk stratification and possibly mitigating the need for biopsies.

DETAILED DESCRIPTION:
Background Prostate cancer (PC) remains a significant cause of morbidity and death among men in Denmark and the rest of the western world. Over 4,500 PC cases are diagnosed every year being the second most common malignancy among men in Denmark. With increasing life expectancy, the incidence of PC is projected to increase. Pivotal to the successful treatment of prostate cancer is establishing an early diagnosis. Localised PC is potentially curable and current curative treatment options have shown efficacy in reducing cancer related mortality.

TRUS biopsies:

Transrectal ultrasound guided prostate biopsies (TRUS biopsies) are conducted routinely for histopathological confirmation in cases of suspected PC. Indication for prostate biopsies include elevated Prostate Specific Antigen (PSA) levels or palpable tumour on digital rectal examination. TRUS biopsies is associated with morbidity in the form of infection, haematuria, rectal bleeding and discomfort. Some of these complications may require hospital admission and can be life threatening.

Current standard biopsy regimes include 10 to 14 systemic biopsy cores taken from the peripheral zone of the prostate. The majority of PC involve the posterior peripheral zone of the prostate readily available for biopsies. The remaining PC are isolated to the transition-, central- and anterior zone of the prostate which are not routinely biopsied on systemic biopsies. Thus, anteriorly located cancers may not be sampled with routine investigations and TRUS biopsies may yield false negative results. As the biopsies are taken randomly throughout the gland, significant cancers located in the peripheral zone will in some cases be missed.

Biomarkers and liquid biopsies:

PSA testing has been widely adopted and more cancers are being detected in Denmark due to unsystematic screening with PSA. PSA is a glycoprotein of the human kallikrein family, and elevated serum concentrations are associated to PC. It is organ specific but not cancer specific, therefore other causes may elevate values, including benign prostatic hyperplasia, prostatitis, urinary tract infections and bladder outlet obstruction. To distinguish prostate cancer from other causes of PSA elevation and to confirm the diagnosis, TRUS biopsies are currently the standard diagnostic test.

A range of novel biomarkers has been proposed to overcome the limitations of PSA's low specificity. Few of these biomarkers have been implemented in clinical practise. In a recently published study, Albitar et al, using a panel of urine and plasma biomarkers, where able to predict biopsy outcomes with a positive predictive value of 90% and negative predictive value of 89% tolerating some low grade cancers (Gleason score < 7). This idea has been disseminated as liquid biopsies.

mpMRI of the prostate: Multiparametric magnetic resonance imaging (mpMRI) of the prostate has emerged as a new technology with the ability to detect PC. Especially in the setting of previously negative TRUS biopsies, mpMRI can provide important additional information enabling targeting of biopsies towards suspected PC lesions. Nevertheless, a PC negative mpMRI may fail to detect cancers in 43% of cases and miss 16% of PCs classified as clinical significant. Thus a negative mpMRI will currently still mandate systemic biopsies. Therefore, novel approaches are needed to better direct biopsies and select patient for biopsies.

Aim

The aim of the current project is to study the following issues:

Assessing the value of prebiopsy mpMRI combined with liquid biopsies in biopsy naive men in predicting biopsy results and possible deriving a diagnostic predictive model.

Assessment of the performance of TRUS mpMRI fusion guided biopsies vs. systemic biopsies combined with liquid biopsies.

Confirming the value of liquid biopsies and investigating its relation to tumour grade and volume.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed written consent.
2. PSA < 20.
3. Referred for prostate biopsy.

Exclusion Criteria::

1. Previously diagnosed with prostate cancer.
2. Active use of anticoagulant (excluding platelet inhibitors) or other contraindication for prostate biopsies.
3. Previously undergone prostate biopsies.
4. Inability to undergo mpMRI scan (pacemaker , claustrophobia, impaired renal function, allergy towards contrast agent etc)
5. Any, previous or current, therapy for benign prostate hyperplasia including surgery or medical therapy (except alpha adrenal blockers).
6. They withdraw their consent.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients will require a prostate, so genotypic gender is a requirement.
Enrollment: 261 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Detection of clinical significant cancer. | 1 month
  Positive biopsies with a Gleason grade > 7.

SECONDARY OUTCOMES:
Detection rate of any cancers | 1 month
  Positive biopsies, any Gleason grade.

OTHER OUTCOMES:
Change in Health Related Quality of Life | Baseline, 24 hour, 1 month and 12 months
  Assessed utilizing the EuroQoL EQ-5D-5L questionnaire (comprising 5 questions with a score from 1 to 5 each and a visual analogue scale from 0 to 100).

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lund, DMsc, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nye kræfttilfælde Tabel [Internet]. Danish Cancer Registry - eSundhed. 2016
- [Background] Bill-Axelson A, Holmberg L, Garmo H, Rider JR, Taari K, Busch C, Nordling S, Haggman M, Andersson SO, Spangberg A, Andren O, Palmgren J, Steineck G, Adami HO, Johansson JE. Radical prostatectomy or watchful waiting in early prostate cancer. N Engl J Med. 2014 Mar 6;370(10):932-42. doi: 10.1056/NEJMoa1311593. PMID 24597866
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Background] Pelzer AE, Bektic J, Berger AP, Halpern EJ, Koppelstatter F, Klauser A, Rehder P, Horninger W, Bartsch G, Frauscher F. Are transition zone biopsies still necessary to improve prostate cancer detection? Results from the tyrol screening project. Eur Urol. 2005 Dec;48(6):916-21; discussion 921. doi: 10.1016/j.eururo.2005.07.012. Epub 2005 Aug 10. PMID 16126324
- [Background] Stamey TA, Yang N, Hay AR, McNeal JE, Freiha FS, Redwine E. Prostate-specific antigen as a serum marker for adenocarcinoma of the prostate. N Engl J Med. 1987 Oct 8;317(15):909-16. doi: 10.1056/NEJM198710083171501. PMID 2442609
- [Background] Albitar M, Ma W, Lund L, Albitar F, Diep K, Fritsche HA, Shore N. Predicting Prostate Biopsy Results Using a Panel of Plasma and Urine Biomarkers Combined in a Scoring System. J Cancer. 2016 Feb 2;7(3):297-303. doi: 10.7150/jca.12771. eCollection 2016. PMID 26918043
- [Background] Panebianco V, Barchetti F, Sciarra A, Ciardi A, Indino EL, Papalia R, Gallucci M, Tombolini V, Gentile V, Catalano C. Multiparametric magnetic resonance imaging vs. standard care in men being evaluated for prostate cancer: a randomized study. Urol Oncol. 2015 Jan;33(1):17.e1-17.e7. doi: 10.1016/j.urolonc.2014.09.013. Epub 2014 Nov 11. PMID 25443268
- [Background] Turkbey B, Pinto PA, Mani H, Bernardo M, Pang Y, McKinney YL, Khurana K, Ravizzini GC, Albert PS, Merino MJ, Choyke PL. Prostate cancer: value of multiparametric MR imaging at 3 T for detection--histopathologic correlation. Radiology. 2010 Apr;255(1):89-99. doi: 10.1148/radiol.09090475. PMID 20308447
- [Background] Boesen L, Noergaard N, Chabanova E, Logager V, Balslev I, Mikines K, Thomsen HS. Early experience with multiparametric magnetic resonance imaging-targeted biopsies under visual transrectal ultrasound guidance in patients suspicious for prostate cancer undergoing repeated biopsy. Scand J Urol. 2015 Feb;49(1):25-34. doi: 10.3109/21681805.2014.925497. Epub 2014 Jun 12. PMID 24922550
- [Background] Filson CP, Natarajan S, Margolis DJ, Huang J, Lieu P, Dorey FJ, Reiter RE, Marks LS. Prostate cancer detection with magnetic resonance-ultrasound fusion biopsy: The role of systematic and targeted biopsies. Cancer. 2016 Mar 15;122(6):884-92. doi: 10.1002/cncr.29874. Epub 2016 Jan 7. PMID 26749141
- [Background] Lamb BW, Tan WS, Rehman A, Nessa A, Cohen D, O'Neil J, Green JS, Hines JE. Is Prebiopsy MRI Good Enough to Avoid Prostate Biopsy? A Cohort Study Over a 1-Year Period. Clin Genitourin Cancer. 2015 Dec;13(6):512-7. doi: 10.1016/j.clgc.2015.06.007. Epub 2015 Jun 30. PMID 26231912